CLINICAL TRIAL: NCT00031720
Title: Phase II Study of Soy Protein to Treat Vasomotor Symptoms in Postmenopausal Women Taking Tamoxifen
Brief Title: Soy Protein Supplement In Treating Hot Flashes in Postmenopausal Women Receiving Tamoxifen for Breast Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Protein Technologies International (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CALGB-79805; U10CA076001 (NIH); CALGB-79805; NCI-P02-0206; CDR0000069219 (Registry Identifier: NCI Physicians Data Query)
Record Dates: First submitted 2002-03-08; First posted 2003-01-27 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Breast Cancer; Hot Flashes; Hot Flushes
Keywords: lobular breast carcinoma in situ; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; recurrent breast cancer; ductal breast carcinoma in situ; hot flashes
MeSH Terms: conditions — Breast Neoplasms; Hot Flashes; Breast Carcinoma In Situ; Carcinoma, Intraductal, Noninfiltrating | interventions — Soybean Proteins; Isoflavones; Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): All patients receive placebo for 7 days as part of the run-in period. Patients being treated with tamoxifen were randomized to treatment arm I and received 40 gm soy protein and 90 mg isoflavones daily for 12 weeks.
  Interventions: Dietary Supplement: soy protein; Dietary Supplement: isoflavones; Drug: Tamoxifen
- Arm II (Placebo Comparator): All patients receive placebo for a 7 day run in period. Patients being treated with tamoxifen randomized to Arm II received placebo daily for 12 weeks.
  Interventions: Drug: Tamoxifen; Other: Placebo

INTERVENTIONS:
Dietary Supplement: soy protein — Given orally
  Arms: Arm I
Dietary Supplement: isoflavones — Given orally
  Arms: Arm I
Drug: Tamoxifen
Other: Placebo — Oral
  Arms: Arm II

SUMMARY:
RATIONALE: Soy protein supplement may be effective in reducing hot flushes in postmenopausal women who are receiving tamoxifen for breast disease.

PURPOSE: Randomized phase II trial to determine the effectiveness of soy protein supplement in reducing hot flushes in postmenopausal women who are receiving tamoxifen for breast disease such as ductal hyperplasia or breast cancer.

DETAILED DESCRIPTION:
OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to duration of hot flashes (less than 9 months vs 9 months or more) and frequency of hot flashes (7 to 9 per day vs more than 9 per day). For more information regarding the treatment regimens, please see the treatment arms section.

Primary objectives:

1. To compare the effect of daily soy supplementation versus placebo on the daily number of hot flushes experienced by postmenopausal women taking tamoxifen measured at three months from baseline
2. To compare the effect of daily soy supplementation versus placebo on hot flush severity as measured by the average daily hot flash score in this population of women measured at three months from baseline

Secondary objectives:

1. To evaluate the effect of soy supplementation as compared to women randomized to placebo on quality of life as measured by the Medical Outcomes Study (MOS) sleep subscale, the Mental Health Inventory (MHI), the CES-D Short Form, the Menopause and Reproductive Health Questionnaire, and the General Quality of Life Form
2. To measure the effect of soy supplementation as compared to women randomized to placebo on serum isoflavones, estradiol, SHBG, IGF1 and IGFBP3 levels as measures of hormonal change
3. To estimate the effect of daily soy supplementation versus placebo on the time to first relief of hot flushes

A total of 112 patients accrued on this study. Patients were followed 6 months post-randomization.

ELIGIBILITY:
Eligibility Criteria:

1. Histologic documentation of atypical ductal hyperplasia, ductal carcinoma in situ (DCIS), lobular carcinoma in situ (LCIS), or invasive adenocarcinoma of the breast stages I-III A.
2. Current daily tamoxifen use. Any planned surgery, adjuvant chemotherapy or radiation must have been completed.
3. History of bothersome hot flushes: ≥ 7 hot flushes/day, sufficiently severe that intervention is desired. Participants must have had bothersome hot flushes for at least one month prior to enrollment.
4. Postmenopausal status: surgical menopause, no menses for ≥ 1 year or postmenopausal FSH levels.
5. No concurrent use of vitamin E, progestins (Megace® or others), clonidine, belladonna derivative or commercially available soy supplement preparations for treatment of hot flushes. Participants must have at least a 4-week washout period prior to day 1 of run-in if any of these have been used.

   Participants may be taking low doses of vitamin E that are part of a multivitamin.
6. Concurrent use of anti-depressant, such as Paxil® , Prozac®, or Effexor® is allowed if the participant has been on a stable dose for more than a month and the purpose of the medication is for other than control of hot flushes. If SSRI's are used for hot flashes, they must be discontinued for 4 weeks prior to day 1 of run-in.
7. No concurrent systemic hormone replacement therapy or use of vaginal estrogen creams. Use of the estradiol releasing vaginal ring (Estring®) is allowed.
8. No history of soy or milk intolerance
9. CALGB performance status 0-2

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2002-03; Primary Completion 2006-04 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Change in number of daily hot flushes at 3 months from baseline | Up to 3 months
Change in hot-flush score at 3 months from baseline | Up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Gini F. Fleming, MD, Study Chair — University of Chicago
Locations (14):
- United States (14):
  - Center for Cancer Care at OSF Saint Anthony Medical Center, Rockford, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - Commonwealth Hematology-Oncology, PC - Worcester, Worcester, Massachusetts
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Kingsbury Center for Cancer Care at Cheshire Medical Center, Keene, New Hampshire
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - FirstHealth Moore Regional Community Hospital Comprehensive Cancer Center, Pinehurst, North Carolina